CLINICAL TRIAL: NCT06840639
Title: The Impact of Dental Health on Complications During and Following Radiotherapy in the Head and Neck Region.
Status: Completed | Type: Observational
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LundUH2
Record Dates: First submitted 2024-11-08; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Neoplasms; Radiotherapy; Complications; Extracting Own Teeth
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Dental extractions with complications: patients recieving dental extractions and developing osteoradionecrosis
  Interventions: Procedure: Dentoalveolar surgery
- Dental extractions without complications: patients recieving dental extractions and not developing osteoradionecrosis

INTERVENTIONS:
Procedure: Dentoalveolar surgery — Surgery to extract teeth
  Groups: Dental extractions with complications

SUMMARY:
Study the risk of complications after dental extractions in patients recieving radiotherapy.

DETAILED DESCRIPTION:
Dental extractions before radiotherapy in the head and neck region is an established part of the treatment plan for patients with malignant disease. There are contradictory results in the literature regarding the importance timing and magnitude of extractions. It is important to minimize complications in this patient group since the regular therapy is already detrimental to the affected tissues. Patients were extracted from the ARTSCAN register were the population was followed for 4 years for several factors, including development of osteoradionecrosis. The aim is to evaluate which diagnoses are more prone to develop complications after extraction. If there is a relationship between occurrence of complication and magnitude of dental pathology.

ELIGIBILITY:
Inclusion Criteria:

* Malignant diagnosis
* radiotherapy pre or postoperative

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients receiving radiotherapy for malignant diagnosis (oral and oropharyngeal cancers)
Sampling Method: Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Does dental extractions increase the risk for complications such as osteoradionecrosis? | From diagnosis of head and neck pathology, approximately 1 month before start of radiotherapy, and to the end of the medical record which may be from one year after the oncologic treatment up to 26 years after oncologic treatment.
  Type of complication when extracting teeth in conjunction with radiotherapy.
Does dental pathology in extracted teeth correlate with development of osteoradionecrosis? | From diagnosis of head and neck pathology, approximately 1 month before start of radiotherapy, and to the end of the medical record which may be from one year after the oncologic treatment up to 26 years after oncologic treatment.
  Are any specific dental pathology more prone to develop complications than others?

CONTACTS AND LOCATIONS:
Overall Officials: Philip Fransson, Msc, Principal Investigator — Lund University Hospital
Locations (1):
- Oral and Maxillofacial department, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided